CLINICAL TRIAL: NCT06827574
Title: Comparative Effects of Sciatic Nerve Flossing and Active Release Technique on Pain, Flexibility and Functionality in Lower Limbs Among Cyclists With Sciatica
Brief Title: Comparative Effects of Sciatic Nerve Flossing and Active Release Technique in Cyclists With Sciatica
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0404
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cyclists; Sciatica
Keywords: Active release technique; cyclists; functional performance; pain management; sciatica; sciatic nerve flossing technique
MeSH Terms: conditions — Sciatica; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sciatic nerve flossing technique (Experimental): Group A 16 subjects were treated with Sciatic Nerve Flossing Technique.
  Interventions: Other: Sciatic nerve flossing technique
- Active Release Technique (Active Comparator): Group B 16 subjects were treated with Active Release Technique
  Interventions: Other: Active Release Technique

INTERVENTIONS:
Other: Sciatic nerve flossing technique — Group A 16 subjects were treated with Sciatic Nerve Flossing Technique. Subjects were in sitting position. Nerve Flossing Technique was performed actively with the participant sitting on a chair. The participant was flex the knee of the target lower extremity backwards beside the chair, as far back as possible and flex the neck at the same time, holding both the flexed knee and neck in this position for 10 seconds. The participant in turn will extend the neck and the knee of the target lower extremity, abduct and then flex the hip until pain is felt and do not push beyond that point. This extended position was maintained for 10 seconds. The above procedure of Nerve Flossing Technique was repeated for 15 times, 3 sets with an interval of 5 minutes between each set. As the nerve becomes less sensitive, the participant can increase the stretching effect by dorsiflexion the ankle and extending the toes of the foot upward towards the shin.
  Arms: Sciatic nerve flossing technique
Other: Active Release Technique — Group B 16 subjects were treated with Active Release Technique. Subjects were in prone position. ART was performed actively by the participant lying on a bed. The participant was dorsiflex the foot of the target lower extremity, holding the dorsiflexion foot in this position for 10 seconds. The participant in turn was plantar-flexed the foot of the target lower extremity. This dorsiflexion position was maintained for 10 seconds. The above procedure of Active Release Technique was repeated for 15 times, 3 sets with an interval of 5 minutes between each set. As the muscles becomes more flexible, the participant can increase the flexibility effect by plantar flexing the foot.
  Arms: Active Release Technique

SUMMARY:
Thus the aim of my study is to determine the comparative effects of sciatic nerve flossing and active release technique on pain, flexibility, and functionality in lower limbs of cyclists with sciatica.

DETAILED DESCRIPTION:
This study investigates the comparative effects of Sciatic Nerve Flossing and Active Release Technique on pain, flexibility, and functionality in cyclists with sciatica. To compare the efficacy of Sciatic Nerve Flossing and Active Release Technique in reducing pain and improving functional performance in cyclists diagnosed with sciatica over a six-week period. A randomized clinical trial was conducted with 32 participants, aged 18 to 35, diagnosed with sciatica persisting for more than six weeks. Participants were randomly assigned to two groups: Group A received Sciatic Nerve Flossing, while Group B underwent Active Release Technique. Pain levels were measured using the Numeric Pain Rating Scale (NPRS), functional performance was assessed using the Lower Extremity Functional Score (LEFS), and flexibility was evaluated via the Sit and Reach Test.

ELIGIBILITY:
Inclusion Criteria

* Age between 18 to 30 years (16)
* Only male participants were included (15)
* Participates with Positive Passive Straight Leg Raise (PSLR) Test (13)
* Athletes with positive slump test (15)
* Symptoms more than 6 weeks (16)

Exclusion Criteria:

* Lower limb fracture(13)
* Musculoskeletal problems (radiculopathy, myopathy) (13, 14)
* Sciatica along with vascular disorders and diabetic neuropathy, sciatica due to tumor and fractures (15)
* Inflammatory arthritis (16)
* Previous surgical interventions on the lower limbs or spine (15)
* Neurological conditions affecting lower limb function (e.g., multiple sclerosis, spinal cord injuries) (13, 14)
* Patients currently undergoing physical therapy or other interventions for sciatica (15)
* Individuals with contraindications to physical activity or exercise due to health conditions (13, 14)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants were included
Enrollment: 32 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
NPRS | 6 Weeks
  The Numeric Aggravation Rating Scale (NPRS) is normally used to survey torment. Change in the NPRS across time can be deciphered with responsiveness lists. Patient level of pain will be assessed using this scale. This scale ranges from 0 to 10. 0 indicates "no pain" and 10 indicates "worst pain(48). High test-retest reliability is indicated by an ICC > 0.70; Cronbach's alpha > 0.70 suggests great internal consistency. The construct validity of the NPRS examines how well the scores correspond to theoretical pain components, while the criterion validity compares results to established pain measures.(49).
Sit and Reach Test | 6 weeks
  Sit-and-arrive at tests are generally utilized as estimation apparatuses for assessing hamstring and lower back adaptability. The old style sits and arrive at test (SRT), initially planned by Wells and Dillon (1952) is frequently included as a feature of game related actual wellness test batteries (American Union for Wellbeing Actual Instruction Entertainment and Dance (AAHPERD), 1986, Gathering of Europe Council for the Improvement of Game, 1993) to assess hamstring muscle adaptability. The SRT and TT test have a similar testing strategy (maximal trunk flexion with knee straight and lower leg in 90° of dorsiflexion) with the main contrast being the trying position, sitting and standing, separately(50).
Lower Extremity Funtional Score | 6 weeks
  The reasonable structure that directed the improvement of the LEFS incorporated that the scale be founded on the World Wellbeing Association's model of incapacity and impairment, be effective to manage, score, and record in the clinical record as for patient and clinician time, be pertinent to a wide assortment of patients with lower-limit muscular circumstances, incorporating patients with a scope of handicap levels, conditions, illnesses, medicines, and ages, be material for reporting capability on a singular patient premise as well as in gatherings, for example, for clinical results evaluation and clinical examination designs, be created utilizing an efficient course of thing determination and thing scaling, yield solid estimations (have inner consistency and test-retest dependability), and yield substantial estimations (at a solitary moment and delicate to legitimate change)(51)(52). While ICC > 0.70 indicates good reliability for LEFS, Cronbach's alpha > 0.70 ensures internal con

CONTACTS AND LOCATIONS:
Overall Officials: Farwa Imtiaz Ahmad, DPT, Principal Investigator — Riphah International University
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiaramonte R, Pavone P, Vecchio M. Diagnosis, Rehabilitation and Preventive Strategies for Pudendal Neuropathy in Cyclists, A Systematic Review. J Funct Morphol Kinesiol. 2021 May 10;6(2):42. doi: 10.3390/jfmk6020042. PMID 34068471
- [Background] Battista S, Sansone LG, Testa M. Prevalence, Characteristics, Association Factors of and Management Strategies for Low Back Pain Among Italian Amateur Cyclists: an Observational Cross-Sectional Study. Sports Med Open. 2021 Oct 28;7(1):78. doi: 10.1186/s40798-021-00370-2. PMID 34709475
- [Background] Zhang YH, Hu HY, Xiong YC, Peng C, Hu L, Kong YZ, Wang YL, Guo JB, Bi S, Li TS, Ao LJ, Wang CH, Bai YL, Fang L, Ma C, Liao LR, Liu H, Zhu Y, Zhang ZJ, Liu CL, Fang GE, Wang XQ. Exercise for Neuropathic Pain: A Systematic Review and Expert Consensus. Front Med (Lausanne). 2021 Nov 24;8:756940. doi: 10.3389/fmed.2021.756940. eCollection 2021. PMID 34901069
- [Background] Chang TT, Li Z, Zhu YC, Wang XQ, Zhang ZJ. Effects of Self-Myofascial Release Using a Foam Roller on the Stiffness of the Gastrocnemius-Achilles Tendon Complex and Ankle Dorsiflexion Range of Motion. Front Physiol. 2021 Sep 17;12:718827. doi: 10.3389/fphys.2021.718827. eCollection 2021. PMID 34603078
- [Background] Mehta SP, Fulton A, Quach C, Thistle M, Toledo C, Evans NA. Measurement Properties of the Lower Extremity Functional Scale: A Systematic Review. J Orthop Sports Phys Ther. 2016 Mar;46(3):200-16. doi: 10.2519/jospt.2016.6165. Epub 2016 Jan 26. PMID 26813750
- [Background] Dingemans SA, Kleipool SC, Mulders MAM, Winkelhagen J, Schep NWL, Goslings JC, Schepers T. Normative data for the lower extremity functional scale (LEFS). Acta Orthop. 2017 Aug;88(4):422-426. doi: 10.1080/17453674.2017.1309886. Epub 2017 Mar 28. PMID 28350206
- [Background] Michener LA, Snyder AR, Leggin BG. Responsiveness of the numeric pain rating scale in patients with shoulder pain and the effect of surgical status. J Sport Rehabil. 2011 Feb;20(1):115-28. doi: 10.1123/jsr.20.1.115. PMID 21411827
- [Background] Danazumi MS, Nuhu JM, Ibrahim SU, Falke MA, Rufai SA, Abdu UG, Adamu IA, Usman MH, Daniel Frederic A, Yakasai AM. Effects of spinal manipulation or mobilization as an adjunct to neurodynamic mobilization for lumbar disc herniation with radiculopathy: a randomized clinical trial. J Man Manip Ther. 2023 Dec;31(6):408-420. doi: 10.1080/10669817.2023.2192975. Epub 2023 Mar 22. PMID 36950742
- [Background] Ashbrook J, Rogdakis N, Callaghan MJ, Yeowell G, Goodwin PC. The therapeutic management of back pain with and without sciatica in the emergency department: a systematic review. Physiotherapy. 2020 Dec;109:13-32. doi: 10.1016/j.physio.2020.07.005. Epub 2020 Jul 23. PMID 32846282
- [Background] Albert HB, Manniche C. The efficacy of systematic active conservative treatment for patients with severe sciatica: a single-blind, randomized, clinical, controlled trial. Spine (Phila Pa 1976). 2012 Apr 1;37(7):531-42. doi: 10.1097/BRS.0b013e31821ace7f. PMID 21494193